CLINICAL TRIAL: NCT04080297
Title: A Two Dose, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Effect on Vasomotor Symptoms of Q-122 in Female Subjects With Breast Cancer and Receiving an Aromatase Inhibitor or Tamoxifen
Brief Title: Dose Escalation Study in Female Subjects With Breast Cancer Receiving Aromatase Inhibitor or Tamoxifen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Que Oncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Q-1001
Record Dates: First submitted 2019-08-20; First posted 2019-09-06 (Actual); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Vasomotor Symptoms (VMS)
Keywords: Vasomotor Symptoms, Breast Cancer, Hot Flashes, Tamoxifen, Aromatase Inhibitors, Estrogen Antagonists, Hormone Antagonists, Hormones, Hormone Substitutes; Hormone Antagonists, Physiological Effects of Drugs, Antineoplastic Agents, Hormonal Antineoplastic, Selective Estrogen Receptor Modulators; Estrogen Receptor Modulators, Bone Density Conservation Agents, Steroid Synthesis Inhibitors, Enzyme Inhibitors, Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes | interventions — N,N'-(1,4-phenylenebis(methylene))dipyrimidin-2-amine

STUDY DESIGN:
Intervention Model Description: open-label, two dose study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 100 mg Q-122 (Experimental): 10 patients treated with Q-122, 100 mg. Dosage was 100 mg Q-122 administered orally as two 50 mg capsules once daily for 28 days.
  Interventions: Drug: oral capsule of Q-122
- 200 mg Q-122 (Experimental): 11 patients treated with Q-122, 200 mg. Dosage was 200 mg Q-122 administered orally as four 50 mg capsules once daily for 28 days.
  Interventions: Drug: oral capsule of Q-122

INTERVENTIONS:
Drug: oral capsule of Q-122

SUMMARY:
Open-label, two dose study of Q-122, over a 4 week treatment period to explore the effects of Q-122 in a population of women with a history of breast cancer taking an aromatase inhibitor or tamoxifen.

DETAILED DESCRIPTION:
Vasomotor symptoms are significant in postmenopausal women with the most effective medications for relief being hormonal preparations. Non-hormonal medications have demonstrated efficacy but at a far lower level than estrogen replacement therapy. For women with a history of breast cancer hormone replacement therapy is problematic especially if their therapeutic regime involves an aromatase inhibitor. Therefore, this study will explore the effect of Q-122 in a population of women with a history of breast cancer taking an aromatase inhibitor or tamoxifen.

The study is an open-label, two dose study (Group 1: 100 mg once daily and Group 2: 200 mg once daily) of Q-122, over a 4 week treatment period. As eligible subjects are enrolled, they will be assigned to Group 1 until Group 1 is fully enrolled. Dose escalation to the 200 mg level will only occur following a review of the safety experience of at least 6 subjects treated with 100 mg Q-122 once daily for at least 2 weeks. Once Group 1 is fully enrolled, eligible subjects will be enrolled into Group 2.

A two-week screening phase will be used to establish a stable baseline of vasomotor symptoms and to establish study eligibility. Qualified subjects will be treated with Q-122 for four weeks either at 100 mg/day dose or the 200 mg/day dose, during which time they will be evaluated for safety, tolerability, and pharmacokinetics of Q-122 and tamoxifen levels; subjects will continue to record their hot flashes in identical fashion to the screening period. Following the 28 day treatment, period subjects who complete the study will continue to record their hot flashes for a two week follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Be a female of any race between the ages of 30-70 years.
* History of breast cancer and presently taking an aromatase inhibitor or tamoxifen.
* Naturally menopausal: ≥ 12 months spontaneous amenorrhea or > 6 but < 12 months amenorrhea with a serum follicle stimulating hormone (FSH) level of > 40 mIU/mL (Milli-international Units Per Milliliter).
* Surgically menopausal with an FSH level > 40 mIU/mL.
* Have a minimum of 7 moderate to severe hot flushes/day or 50 moderate to severe hot flushes per week, as verified for both weeks during the 14-day Screening Phase, prior to enrollment into the treatment phase of the study.
* Able to read, understand and complete the required subject diary.
* Willing and able to complete the daily subject diary, attend all study visits, and participate in all study procedures, including PK blood draws.

Exclusion Criteria:

* Childbearing potential, including pregnancy, or lactation.
* Undiagnosed abnormal genital bleeding.
* Significant day-to-day variability in hot flushes.
* Participation in another clinical trial within 30 days prior to screening or during the study.
* Legal incapacity or limited legal capacity.
* Chronic renal (serum creatinine > 2.0 mg/dL) or hepatic disease [SGPT (ALT) or SGOT (AST) > 2X normal limits].
* Gastrointestinal, liver, kidney or other conditions which could interfere with the absorption, distribution, metabolism or excretion of Q-122.
* Untreated overt hyperthyroidism.
* Use of thyroid medication of less than 12 weeks on a stable dose.
* Any clinically important systemic disease in the judgement of the investigator.
* Inability to complete all study visits and study assessments for scheduling or other reasons.
* Any other reason which in the investigator's opinion makes the subject unsuitable for a clinical trial.
* Abnormal laboratory findings including:

  1. Hematocrit < 30% or hemoglobin < 9.5 gm/dL
  2. Fasting blood sugar > 140 mg/dL
  3. Fasting serum triglycerides > 300 mg/dL
  4. Fasting SGOT, SGPT, GGT, or bilirubin greater than twice the upper limit of normal (a subject will not be excluded if a second measurement is less than twice the upper limit of normal)
  5. Creatinine > 2.0 mg/dL

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 21 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2014-07-28 (Actual); Study Completion 2014-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rob Crombie, Study Chair — Que Oncology

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- 100 mg Q-122: Dosage was 100 mg Q-122 administered orally as two 50 mg capsules once daily for 28 days.
- 200 mg Q-122: Dosage was 200 mg Q-122 administered orally as four 50 mg capsules once daily for 28 days.
Period: Overall Study
Arm/Group | 100 mg Q-122 | 200 mg Q-122
Started | 10 | 11
Completed | 8 | 8
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 3
Not completed — concurrent illness | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 mg Q-122 | 200 mg Q-122 | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Median (Full Range); unit: years] | 56.5 [48 to 64] | 57 [47 to 67] | 56.8 [47 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 9 | 19
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Adverse Event (AE) Reporting of Q-122
Description: Number of participants with indicated AE receiving Q-122
Time Frame: 4 weeks
Population: Analyses were performed using the results from the safety analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | 100 mg Q-122 | 200 mg Q-122
Number analyzed (Participants) | 10 | 11
Participants | 7 | 7

2. Primary Outcome: Serious Adverse Event (SAE) Reporting of Q-122
Description: Number of participants with indicated SAE receiving Q-122
Time Frame: 4 weeks
Population: Analyses were performed using the results from the safety analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | 100 mg Q-122 | 200 mg Q-122
Number analyzed (Participants) | 10 | 11
Participants | 0 | 1

3. Primary Outcome: Change in Frequency of Moderate to Severe Vasomotor Symptoms.
Description: Mean change in frequency of moderate to severe vasomotor symptoms. Daily patient (paper) diaries will be used as the primary efficacy collection tool. Change from baseline represents the mean change from the daily average frequency calculated at baseline to the daily average frequency calculated for the last week the subject was on drug. The hot flash severity categories are defined clinically as follow: mild, sensation of heat without perspiration; moderate, sensation of heat with perspiration, but subject is able to continue with activity; and severe. sensation of heat with sweating, sufficiently severe to result in discontinuation of activity.
Time Frame: Baseline to 4 weeks
Population: Analyses were performed using the intent-to-treat (ITT) population.
Measure: Mean (Standard Deviation); unit: Hot flashes/day
Arm/Group | 100 mg Q-122 | 200 mg Q-122
Number analyzed (Participants) | 10 | 11
Hot flashes/day
  Baseline: number analyzed (Participants) | 9 | 11
  Baseline | 9.86 (3.18) | 8.58 (1.63)
  Change from baseline: number analyzed (Participants) | 8 | 8
  Change from baseline | -5.81 (3.71) | -5.60 (3.13)

4. Primary Outcome: Percent Change in Frequency of Moderate to Severe Vasomotor Symptoms.
Description: Percent reduction in frequency of moderate to severe vasomotor symptoms. Daily patient (paper) diaries will be used as the primary efficacy collection tool. The hot flash severity categories are defined clinically as follows: mild, sensation of heat without perspiration; moderate, sensation of heat with perspiration, but subject is able to continue with activity; and severe, sensation of heat with sweating, sufficiently severe to result in discontinuation of activity.
Time Frame: Baseline to 4 weeks
Population: Analyses were performed using the intent-to-treat (ITT) population.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 100 mg Q-122 | 200 mg Q-122
Number analyzed (Participants) | 9 | 11
Percent change | -61.46 (38.85) | -67.55 (39.27)

5. Secondary Outcome: Change in Hot Flash Severity Score
Description: For moderate-to-severe (mod/sev) hot flashes (HF), a score will be calculated by multiplying the number of moderate-to-severe HFs by their severity to determine the HF (mod/sev) index score, using the following formula: HFSSmod/sev = (number of moderate hot flashes/day × 2) + (number of severe hot flashes/day x 3). The Average Daily HFSSmod/sev for each week will be calculated by dividing the total of daily HFSSmod/sev by the number of days observations will be recorded in that week. The change in score is of clinical significance, with a lower score representing less moderate to severe hot flashes and a higher score representing a greater number of moderate to severe hot flashes.
Time Frame: Baseline to 4 weeks
Population: Analyses were performed using the intent-to-treat (ITT) population. The ITT population was defined as all subjects who received at least one dose of study medication and have an evaluable primary or secondary efficacy measurement after baseline.
Measure: Mean (Standard Deviation); unit: Hot flash severity score (HFSS)/day
Arm/Group | 100 mg Q-122 | 200 mg Q-122
Number analyzed (Participants) | 10 | 11
Hot flash severity score (HFSS)/day
  Baseline: number analyzed (Participants) | 9 | 11
  Baseline | 24.91 (10.76) | 20.64 (4.06)
  Treatment - Week 1: number analyzed (Participants) | 9 | 11
  Treatment - Week 1 | 17.67 (13.87) | 10.09 (6.74)
  Treatment - Week 2: number analyzed (Participants) | 9 | 10
  Treatment - Week 2 | 12.41 (12.58) | 9.51 (7.41)
  Treatment - Week 3: number analyzed (Participants) | 8 | 10
  Treatment - Week 3 | 10.11 (12.81) | 9.35 (8.73)
  Treatment - Week 4: number analyzed (Participants) | 8 | 8
  Treatment - Week 4 | 11.14 (14.23) | 7.89 (10.06)

6. Secondary Outcome: Percent Change in Hot Flash Severity Score
Description: For moderate-to-severe (mod/sev) hot flashes (HF), a score will be calculated by multiplying the number of moderate-to-severe HFs by their severity to determine the HF (mod/sev) index score, using the following formula: HFSSmod/sev = (number of moderate hot flashes/day × 2) + (number of severe hot flashes/day x 3). The Average Daily HFSSmod/sev for each week will be calculated by dividing the total of daily HFSSmod/sev by the number of days observations will be recorded in that week.
Time Frame: Baseline to 4 weeks
Population: Analyses were performed using the intent-to-treat (ITT) population.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 100 mg Q-122 | 200 mg Q-122
Number analyzed (Participants) | 9 | 11
Percent change | -61.97 (36.03) | -67.55 (40.81)

7. Secondary Outcome: Symptoms Associated With Postmenopausal Status
Description: Greene Climacteric Scale: A comprehensive assessment divided into psychological, physical and vasomotor areas. The scale includes 21 symptoms, subject will score the severity of each symptom with the following score system: 0 = not at all; 1 = a little; 2 = quite a bit; and 3 = extremely. The results represent the total combined score, which can range from 0 to 63. A lower score represents a better outcome.
Time Frame: Baseline and 4 weeks
Population: Analyses were performed using the intent-to-treat (ITT) population. The ITT population was defined as all subjects who received at least one dose of study medication and had an evaluable primary or secondary efficacy measurement after baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 100 mg Q-122 | 200 mg Q-122
Number analyzed (Participants) | 10 | 11
score on a scale
  Total Score - Baseline: number analyzed (Participants) | 9 | 11
  Total Score - Baseline | 18.1 (6.15) | 19.1 (12.38)
  Total Score - 4 weeks: number analyzed (Participants) | 8 | 8
  Total Score - 4 weeks | 6.5 (5.95) | 4.5 (2.88)

ADVERSE EVENTS:
Arm/Group | 100 mg Q-122 | 200 mg Q-122
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/11
Other Adverse Events (participants affected / at risk) | 7/10 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 mg Q-122 (N=10) | 200 mg Q-122 (N=11)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 mg Q-122 (N=10) | 200 mg Q-122 (N=11)
Aspartate aminotransferase increase (Investigations) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (3)
Insomnia (Nervous system disorders) | 0 (0) | 1 (1)
Gastroenteritis viral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral herpes (Gastrointestinal disorders) | 0 (0) | 1 (1)
Contusion (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Euphoric mood (Psychiatric disorders) | 0 (0) | 1 (1)
Flank pain (General disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No